CLINICAL TRIAL: NCT04896528
Title: Efficacy and Safety of Avatrombopag in Cancer Patients With Thrombocytopenia Induced by Targeted Therapy and Immunotherapy Combination Treatment
Brief Title: Efficacy and Safety of Avatrombopag in Cancer Patients With Thrombocytopenia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SKX-CIT-002
Record Dates: First submitted 2021-04-28; First posted 2021-05-21 (Actual); Last update posted 2021-05-21 (Actual); Status verified 2021-04

CONDITIONS: Thrombocytopenia; Avatrombopag
MeSH Terms: conditions — Thrombocytopenia | interventions — avatrombopag

STUDY DESIGN:
Intervention Model Description: Patients receiving combined targeted therapy (including but not limited to tyrosine kinase inhibitors, cyclin-dependent kinase inhibitors) with immunotherapy (including but not limited to PD-1 inhibitors and/or PD-L1 inhibitors and/or CTLA-4 inhibitors); Patients experienced grade III or above thrombocytopenia (PC ≤50×109/L) at least once within 48 h of the screening period;
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Avatrombopag (Experimental): Avartripopa is a new generation of oral TPO receptor agonist that simulates the biological effects of TPO in vitro and in vivo.
  TPO stimulates megakaryocytes through binding and activation of TPO receptor, which is expressed in hematopoietic stem cells, megakaryotic cell lines and platelets.
  By binding to the transmembrane region of the thrombopoietin receptor, Ava Tripopa activates the thrombopoietin receptor in humans, stimulates signal transduction and mimics the biological effects of thrombopoietin, leading to an increase in platelet count.
  Interventions: Drug: Avatrombopag

INTERVENTIONS:
Drug: Avatrombopag — * Participants meeting the eligibility criteria receive Avatrombopag treatment (orally, 60 mg/day), for a maximum course of 20 days.
  * Investigation product withdrawal: PLT ≥75×109/L or increases by at least 50×109/L from the lowest value after targeted therapy and immunotherapy combination treatment.

SUMMARY:
To evaluate the efficacy and safety of Avatrombopag in patients with thrombocytopenia induced by targeted therapy and immunotherapy combination treatment, and provide evidence-based medication for the clinical use of Avatrombopag in patients with PC ≤50×109/L

DETAILED DESCRIPTION:
This phase II trial is a single-arm, non-randomized and single-center clinical study.

It is estimated that 30 patients who met the study criteria will be enrolled in PUMCH and treated with Avatrombopag. The investigators will follow up and collect subjects' data each month to evaluate the efficacy and safety of treatment. Primary outcome measure is percentage of participants whose PLT reaches ≥75×109/L, or increases by ≥50×109/L or ≥100% from baseline at least once within 20 days of initial treatment.

Secondary outcome measure:1)Number of days required for PLT to reach ≥50×109/L after treatment; 2)Number of days required for PLT to reach ≥75×109/L after treatment; 3)Percentage of subjects without platelet transfusion within 20 days of treatment; 4)Percentage of subjects without clinically relevant bleeding within 20 days of treatment.

Study Type: Interventional. Masking: Open Label.

ELIGIBILITY:
Inclusion Criteria:

Each participant must meet all of the following criteria:

1. Male or female, 18~85 years of age;
2. Diagnosis of malignant solid tumor;
3. Participants receiving combined targeted therapy (including but not limited to tyrosine kinase inhibitors, cyclin-dependent kinase inhibitors) with immunotherapy (including but not limited to PD-1 inhibitors and/or PD-L1 inhibitors and/or CTLA-4 inhibitors);
4. Participants experienced grade III or above thrombocytopenia (PC ≤50×109/L) at least once within 48 h of the screening period; No oral platelet-enhancing drugs were given before enrollmen.
5. ECGO performance status ≤2;
6. Blood test:

   * Hemoglobin (Hb) ≥ 9.0 g/dL;
   * Absolute neutrophils count (ANC) ≥ 1,500/μL;
7. Liver and renal functions:

   * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3*ULN (Upper Limits of Normal);
   * Serum bilirubin ≤ 1.5*ULN;
   * Albumin ≥ 2.5 g/dL;
   * Serum creatinine ≤ 1.5*ULN (CTCAE Grade Ⅰ)
8. Participants able to oral medication;
9. Expected survival time ≥12 weeks during screening period;
10. Participants with negative urine or serum pregnancy test during screening period; fertile potential participants must agree to use contraception for the whole study period and 30 days after discontinuity of investigational product treatment (infertile potential was defined as the condition including hysterectomy and bilateral oophorectomy, bilateral salpingectomy, tubal ligation and postmenopausal);
11. Participants in the trial is voluntary and must strictly abide by the protocol;
12. Participants must sign the written informed consent form.

Exclusion Criteria:

Participants meeting any of the following criteria will be excluded from the study:

1. Participants has any history of active congestive heart failure [New York Heart Association (NYHA) Grade III-IV], symptomatic ischemia, uncontrolled arrhythmia, pericardial disease, or myocardial infarction during the first 4 months of enrollment;
2. Participants finished major operation within less than 28 days and for minor operation within less than 3 days;
3. Participants had clinically significant acute or active bleeding (e.g., gastrointestinal or central nervous system) within 7 days prior to screening;
4. Participants has medical-known hereditary prethrombotic syndrome (such as factor V Leiden mutation, prothrombin G20210A mutation or hereditary antithrombin III deficiency);
5. Participants has a history of arterial or venous thrombosis within 3 months prior to screening;
6. Participants had treatment with heparin and warfarin within 7 days prior to screening;
7. Participants has history of chronic thrombocytopenia or hemorrhagic disease, or thrombocytopenia induced by other reasons besides targeted therapy and immunotherapy combination treatment(e.g., chronic liver disease or immune thrombocytopenic purpura);
8. Participants had the treatment of platelet transfusion within 3 days before enrollment;
9. Participants had administration of platelet growth factor (e.g., rhTPO, rhIL-11, Eltrombopag, or Romiplostim) for the treatment of thrombocytopenia induced by targeted therapy and immunotherapy combination treatment within 2 weeks prior to screening;
10. Participants' thrombocytopenia responded effectively to hormone therapy;
11. Participants are allergic to Avatrombopag or any of its excipients;
12. Participants were in any other clinical trial of investigational product or device within 30 days prior to screening, except for observational study;
13. Participants have any known concomitant history that may impair the safe completion of the study as assessed by the investigator, such as unstable angina, renal failure due to hemodialysis, or active infection requiring intravenous antibiotics;
14. Participants are pregnant or lactating at the time of screening (as demonstrated by a positive serum β-HCG test) or baseline visit (positive urine β-HCG test)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-06-06 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants' PLT | one year
  Percentage of participants whose PLT reaches ≥75×109/L, or increases by ≥50×109/L or ≥100% from baseline at least once within 20 days of initial treatment.

SECONDARY OUTCOMES:
Number of days required for PLT to reach ≥50×109/L after treatment; | one year
Number of days required for PLT to reach ≥75×109/L after treatment; | one year
Percentage of subjects without platelet transfusion within 20 days of treatment; | one year
Percentage of subjects without clinically relevant bleeding within 20 days of treatment. | one year

CONTACTS AND LOCATIONS:
Overall Officials: Haitao Haitao, Prof, Study Chair — Peking Union Medical College Hospital (PUMCH)
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arora S, Balasubramaniam S, Zhang W, Zhang L, Sridhara R, Spillman D, Mathai JP, Scott B, Golding SJ, Coory M, Pazdur R, Beaver JA. FDA Approval Summary: Pembrolizumab plus Lenvatinib for Endometrial Carcinoma, a Collaborative International Review under Project Orbis. Clin Cancer Res. 2020 Oct 1;26(19):5062-5067. doi: 10.1158/1078-0432.CCR-19-3979. Epub 2020 Apr 15. PMID 32295834
- [Result] Lingen MW, Kalmar JR, Karrison T, Speight PM. Critical evaluation of diagnostic aids for the detection of oral cancer. Oral Oncol. 2008 Jan;44(1):10-22. doi: 10.1016/j.oraloncology.2007.06.011. Epub 2007 Sep 6. PMID 17825602
- [Result] Adelstein DJ, Li Y, Adams GL, Wagner H Jr, Kish JA, Ensley JF, Schuller DE, Forastiere AA. An intergroup phase III comparison of standard radiation therapy and two schedules of concurrent chemoradiotherapy in patients with unresectable squamous cell head and neck cancer. J Clin Oncol. 2003 Jan 1;21(1):92-8. doi: 10.1200/JCO.2003.01.008. PMID 12506176
- [Result] Pignon JP, le Maitre A, Maillard E, Bourhis J; MACH-NC Collaborative Group. Meta-analysis of chemotherapy in head and neck cancer (MACH-NC): an update on 93 randomised trials and 17,346 patients. Radiother Oncol. 2009 Jul;92(1):4-14. doi: 10.1016/j.radonc.2009.04.014. Epub 2009 May 14. PMID 19446902
- [Result] Suntharalingam M, Haas ML, Conley BA, Egorin MJ, Levy S, Sivasailam S, Herman JM, Jacobs MC, Gray WC, Ord RA, Aisner JA, Van Echo DA. The use of carboplatin and paclitaxel with daily radiotherapy in patients with locally advanced squamous cell carcinomas of the head and neck. Int J Radiat Oncol Biol Phys. 2000 Apr 1;47(1):49-56. doi: 10.1016/s0360-3016(00)00408-9. PMID 10758304
- [Result] Garden AS, Harris J, Vokes EE, Forastiere AA, Ridge JA, Jones C, Horwitz EM, Glisson BS, Nabell L, Cooper JS, Demas W, Gore E. Preliminary results of Radiation Therapy Oncology Group 97-03: a randomized phase ii trial of concurrent radiation and chemotherapy for advanced squamous cell carcinomas of the head and neck. J Clin Oncol. 2004 Jul 15;22(14):2856-64. doi: 10.1200/JCO.2004.12.012. PMID 15254053
- [Result] Adkins D, Ley J, Michel L, Wildes TM, Thorstad W, Gay HA, Daly M, Rich J, Paniello R, Uppaluri R, Jackson R, Trinkaus K, Nussenbaum B. nab-Paclitaxel, cisplatin, and 5-fluorouracil followed by concurrent cisplatin and radiation for head and neck squamous cell carcinoma. Oral Oncol. 2016 Oct;61:1-7. doi: 10.1016/j.oraloncology.2016.07.015. Epub 2016 Jul 29. PMID 27688097
- [Result] Reddy BK, Lokesh V, Vidyasagar MS, Shenoy K, Babu KG, Shenoy A, Naveen T, Joseph B, Bonanthaya R, Nanjundappa, Bapsy PP, Loknatha, Shetty J, Prasad K, Tanvir Pasha CR. Nimotuzumab provides survival benefit to patients with inoperable advanced squamous cell carcinoma of the head and neck: a randomized, open-label, phase IIb, 5-year study in Indian patients. Oral Oncol. 2014 May;50(5):498-505. doi: 10.1016/j.oraloncology.2013.11.008. Epub 2014 Mar 6. PMID 24613543